CLINICAL TRIAL: NCT06454123
Title: A Feasibility Study of a Digital Therapeutic for Adults With Recurrent Binge Eating and Obesity
Brief Title: Feasibility of a Digital Therapeutic for Adults With Binge Eating and Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oui Therapeutics, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-Oui-001; 1R41MH134704-01 (NIH)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Binge Eating; Obesity
MeSH Terms: conditions — Bulimia; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: OTX-401

INTERVENTIONS:
Device: OTX-401 — Evidence-based treatments for obesity and binge eating

SUMMARY:
The primary objective of this study is to test the feasibility of a digital therapeutic to address comorbid binge eating and obesity in adults.

DETAILED DESCRIPTION:
This single-arm, open-label clinical trial will test the feasibility, usability, acceptability, and preliminary efficacy of a digital therapeutic in reducing binge eating and weight in 30 adults with comorbid recurrent binge eating and obesity.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking male or female patients, 18-70 years
2. Patients with recurrent binge eating (≥12 episodes in 3 months) and obesity (BMI ≥30)
3. Understand written and spoken English
4. Own an iPhone with iOS 11 or higher, or Android with OS 8.1 or higher
5. Willing and able to complete enrollment procedures
6. Able to understand the nature of the study and provide written informed consent

Exclusion Criteria:

1. Patients with active psychosis
2. Patients who are acutely intoxicated at the time of enrollment
3. Currently enrolled in other treatment studies for the symptoms and behaviors targeted
4. Patients who are cognitively impaired
5. Patients who, in the judgment of the investigator, would have an unfavorable risk/benefit profile with respect to the digital therapeutic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
System Usability Sale (SUS) | Week 12
  The SUS and a semi-structured user feedback interview will be utilized to systematically capture usability and acceptability.